CLINICAL TRIAL: NCT04098731
Title: Evaluation of Respiratory Function in People With Fibromyalgia
Brief Title: Evaluation of Respiratory Function in Fibromyalgia
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: uppsala18
Record Dates: First submitted 2019-08-20; First posted 2019-09-23 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Fibromyalgia; Respiratory Alkalosis and Metabolic Acidosis; Chronic Hyperventilation
Keywords: Fibromyalgia; Respiratory function
MeSH Terms: conditions — Fibromyalgia; Alkalosis, Respiratory; Acidosis; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will evaluate respiratory function in people with fibromyalgia and whether or not breathing patterns in this patient group can be explained by stress, emotional or biomechanical variables. In addition, examine the relationship between physical ability and lactate values.

DETAILED DESCRIPTION:
Fibromyalgia is characterized by persistent widespread pain and affects approximately 1-3% of the general population. Fibromyalgia is a multifactorial syndrome and much research has been done and several interesting facts discovered. Still, the etiology is unknown. The autonomic nervous system may be the cause of several symptoms of this condition and a pattern of abnormal autonomous functions has been described . Besides the autonomous nerve system the respiratory system has also potential to impact various body organs mainly by altered blood gas chemistry. Deviant respiratory function in local pain condition as in cervical and lumbar spine has been reported. Respiratory function in generalized pain as in people with fibromyalgia has not been given much consideration.

This project is an observational cross sectional study with the purpose to examine respiratory function in people with fibromyalgia and compare with age-matched controls.

Respiratory function will be examined by spirometry and blood gases. Both static (vital capacity, tidal volume) and dynamic lung volumes (forced vital capacity, forced expiratory volume in 1 second) and the ratio of forced expiratory volume in 1 second and forced vital capacity will be used. Spirometry will be performed in seated position. Respiratory rate will be examined in a sitting position using intensive care equipment with electrodes placed under each clavicle and over the lower ribs on the left side. After five minutes of relaxing, breathing frequency is observed during one minute. A value is noted every ten second and a mean value is calculated. Subjects are not aware of when the observation begin. An arterial blood sample will be taken to determine carbon dioxide, oxygen, saturation, bicarbonate, pH and base excess levels. Other blood samples that will be taken is magnesium in venous blood and lactate in capillary blood. Arterial and venous blood samples will be taken in supine position while capillary samples will be done in seated position. Lactate will be sampled before and directly after a six minutes walking test.

Chest mobility, postural balance, spinal mobility, pain sensitivity test and body mass index will be measured as physical or biomechanical variables. By using a tape measure chest mobility will be measured in a standing position at the xiphoid process and axillary level. Spinal mobility will be measured in a seated position between C7-T5 measuring the difference between upright position and full flexion of the spine. By using an analyzing software program called Cervico thoracic ratio 5.0, postural balance can be calculated based on the same method of measuring spinal mobility described above. Pain sensitivity test will be performed over paraspinal muscles between the level of C7-T7 with a total of 14 locations by using a pressure algometer with the subject lying prone. Measurement of the subject's weight and height will be recorded and the body mass index (BMI) will be calculated.

Heart rate variability and self administered questionnaires (Hospital and anxiety depression scale, Pain catastrophizing scale, Perceived stress scale, Montgomery-Asberg Depression Rating Scale) will be used to assess stress or emotional variables. The Rand 36-item will be used as a quality-of-life measurement. Heart rate variability will be measured during five minutes by a portable ECG device in a sitting position with electrodes placed under each clavicle and over the lower ribs on the left side. Questionnaires are encouraged to be filled in before the visit.

For physical function a standardized six minutes walking test and a chair stand test will take place for measuring endurance and strength.

All measurement will be executed at the same visit. Data about smoking habits, pain duration, analgetic drug use will be registered.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with fibromyalgia according to American College of Rheumatology criteria 2010.
* Age 20 to 65 years
* Informed consent.

Exclusion Criteria:

* Trauma in neck-shoulder or thoracic region with prolonged symptoms during the last three months before examination.
* Severe illness (neurological e.g Parkinson disease, neuromuscular e.g Multiple sclerosis, respiratory e.g chronic obstructive pulmonary disease, muscle/skeletal disease e.g ankylosing spondylitis)
* Inability to understand or follow instructions in Swedish
* Use of antidepressant drugs
* For the healthy controls, any other complaints from the chest wall and neck and shoulder region within three month before examination.

N.B Smoking will not be an exclusion criterion.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosed fibromyalgia and healthy subjects included as controls.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in percentage (FEV%) | Day 1
  The forced expiratory volume in percentage will be determined by the ratio of the forced expiratory volume in one second (L/sec) and the forced vital capacity (L). A spirometer is used for these respiratory tests.
Partial pressure of carbon dioxide | Day 1
  An arterial (radial) blood gas test will be performed to measure the carbon dioxide partial pressure (kPa).

SECONDARY OUTCOMES:
Respiratory rate | Day 1
  Respiratory rate is the number of breaths a person take per minute (number per minute). Respiratory rate will be measured by using intensive care equipment. Electrodes will be placed under each clavicle and over the lower ribs on the left side. The equipment sense the distance between the electrodes i.e the movement of the chest wall. After five minutes of relaxing, respiratory rate is measured during one minute.

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Peterson, MD PhD, Principal Investigator — Uppsala University
Locations (1):
- Nyköping hospital, Nyköping, Sörmland, Sweden

REFERENCES:
- [Derived] Jonsson K, Pikwer A, Olsson EM, Peterson M. Altered breathing pattern and thoracic mobility in women with fibromyalgia: A case-control study. J Pain. 2025 Oct;35:105508. doi: 10.1016/j.jpain.2025.105508. Epub 2025 Jul 22. PMID 40706939